CLINICAL TRIAL: NCT04944446
Title: Effectiveness of Myofascial Release in Pathologies of the Shoulder
Brief Title: Myofascial Release in Shoulder Pathologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: InesCarmona
Record Dates: First submitted 2020-09-23; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Humerus Fracture; Rotator Cuff Injuries
Keywords: Shoulder; Pathology; Myofascial release; Clinical trial
MeSH Terms: conditions — Humeral Fractures; Rotator Cuff Injuries | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled longitudinal experimental study
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) external evaluator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group myofascial treatment (Experimental): The trial group will also be referred by the rehabilitating doctor to the physiotherapy room, these patients will be treated by two physiotherapists with training in myofascial release therapy with which they will carry out a treatment protocol that will consist of myofascial release of the shoulder blade angle, subscapularis and global pectoral technique as well as superficial myofascial release of said musculature with a during 12-15 minutes, in addition to a 30-minute session of active kinesitherapy with exercises and mechanotherapy. Same as the control group.
  These mobilizations are carried out in the absence of pain, although the difference between joint tension or stretching and pain is explained to the patient.
  Interventions: Other: Treatment
- Group Kinesitherapy treatment (Active Comparator): This group will be treated in a protocolized way with techniques such as passive kinesitherapy, active-assisted and active kinesitherapy to win mobility.
  They consist of mobilizing the affected arm in the movements of flexion (upward), separation (towards the outer side) and rotation, these lateral decubitus (bring the hand to the nape of the neck) and internal (bring the hand to the lower back) trying to win joint amplitude.
  These mobilizations are performed in the absence of pain, although the difference between joint tension or stretching and pain will be explained to the patient. The treatment will be carried out as usual with a duration of about 12-15 minutes of mobilization and about 30 minutes of active kinesitherapy with exercises and mechanotherapy, these consist of active shoulder mobility exercises. Emphasis will be placed on working with the pain threshold so as not to cause damage or negative nociceptive reactions.
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — Myofascial release of various muscle groups Treatment of mobilization of the shoulder joint

SUMMARY:
Shoulder pathology has a high prevalence in the field of musculoskeletal diagnoses, as well as being a common etiology in cases of disability. Passive and active-assisted kinesitherapy are used in the physiotherapy protocol. These techniques sometimes lead to feedback of fear and increased sensation of pain on the part of the patient that can slow or hinder the optimal recovery. A randomized clinical trial is intended to demonstrate that techniques for myofascial release of muscles important in the biomechanics of the shoulder, it is more effective than kinesitherapy in improving myofascial and also by eliminating the aforementioned unwanted effects and, therefore, improving the recovery of these processes.

DETAILED DESCRIPTION:
The purpose of this study was to compare the efficacy of myofascial therapy and kinesitherapy in improving function in shoulder pathology with prolonged immobilization. Design Prospective, single-blind randomized controlled trial. Setting Inpatient department of a secondary university hospital. Participants Shoulder pain patients (N=44) were consecutively recruited and randomly assigned to an intervention or control group. Interventions Patients were randomly assigned to a Control Group, to which conventional kinesitherapy was applied, or to the intervention group to which a Myofascial therapy protocol was applied. Both groups completed a therapeutic exercise program based on specific mobilization and strengthening exercises. Main Outcome Measures The QuickDash questionnaire was the primary outcome, visual analog scale and the passive range of motion of the shoulder joint, grades were the secondary outcomes. The outcomes were evaluated at baseline (T0) and at 4 (T2),

ELIGIBILITY:
Inclusion Criteria:

* Be between 20 and 80 years old.
* Patients who have been immobilized due to the following diagnoses: Suture of the rotator cuff or fracture of the proximal extremity of the humerus.
* Have signed the informed consent of acceptance in the participation of the study

Exclusion Criteria:

* Present neurological pathology.
* Be subdued corticoid therapy.
* Have anticoagulant treatment or have had it less than a month ago.
* Insulin-dependent diabetic patients.
* Patients with hemophilia.
* Having diagnosed a psychological or psychiatric pathology.
* Non-intervened displaced humerus fractures.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Functional capacity | Baseline
  Dash Scale. Minimum: 0 Maximum: 100. Higher scores mean a worse outcome
Shoulder joint mobility | Baseline
  Goniometer Records
Degree of pain | Baseline
  Visual Analog Scale. Minimum: 0 Maximum: 10. Higher scores mean a worse outcome
Functional capacity | Change from Baseline at 4 weeks
  Dash Scale. Minimum: 0 Maximum: 100. Higher scores mean a worse outcome
Shoulder joint mobility | Change from Baseline at 4 weeks
  Goniometer Records
Degree of pain | Change from Baseline at 4 weeks
  Visual Analog Scale

SECONDARY OUTCOMES:
Pathology of access to the study | Baseline
  Suture of the rotator cuff or fracture of the proximal limb of the humerus
Age | Baseline
  Years
Sex | Baseline
  Man or woman

CONTACTS AND LOCATIONS:
Overall Officials: Inés Carmona Barrientos, Dra., Principal Investigator — University of Cádiz
Locations (1):
- Faculty of Nursing and Physiotherapy. University of Cadiz, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ajimsha MS, Al-Mudahka NR, Al-Madzhar JA. Effectiveness of myofascial release: systematic review of randomized controlled trials. J Bodyw Mov Ther. 2015 Jan;19(1):102-12. doi: 10.1016/j.jbmt.2014.06.001. Epub 2014 Jun 13. PMID 25603749
- [Result] Castro-Martin E, Ortiz-Comino L, Gallart-Aragon T, Esteban-Moreno B, Arroyo-Morales M, Galiano-Castillo N. Myofascial Induction Effects on Neck-Shoulder Pain in Breast Cancer Survivors: Randomized, Single-Blind, Placebo-Controlled Crossover Design. Arch Phys Med Rehabil. 2017 May;98(5):832-840. doi: 10.1016/j.apmr.2016.11.019. Epub 2016 Dec 18. PMID 28003133
- [Result] Rodriguez-Fuentes I, De Toro FJ, Rodriguez-Fuentes G, de Oliveira IM, Meijide-Failde R, Fuentes-Boquete IM. Myofascial Release Therapy in the Treatment of Occupational Mechanical Neck Pain: A Randomized Parallel Group Study. Am J Phys Med Rehabil. 2016 Jul;95(7):507-15. doi: 10.1097/PHM.0000000000000425. PMID 26745225
- [Result] Ajimsha MS, Chithra S, Thulasyammal RP. Effectiveness of myofascial release in the management of lateral epicondylitis in computer professionals. Arch Phys Med Rehabil. 2012 Apr;93(4):604-9. doi: 10.1016/j.apmr.2011.10.012. Epub 2012 Jan 10. PMID 22236639
- [Result] Castro-Sanchez AM, Mataran-Penarrocha GA, Granero-Molina J, Aguilera-Manrique G, Quesada-Rubio JM, Moreno-Lorenzo C. Benefits of massage-myofascial release therapy on pain, anxiety, quality of sleep, depression, and quality of life in patients with fibromyalgia. Evid Based Complement Alternat Med. 2011;2011:561753. doi: 10.1155/2011/561753. Epub 2010 Dec 28. PMID 21234327
- [Derived] Sumariva-Mateos J, Leon-Valenzuela A, Vinolo-Gil MJ, Bautista Troncoso J, Del Pino Algarrada R, Carmona-Barrientos I. Efficacy of myofascial therapy and kinesitherapy in improving function in shoulder pathology with prolonged immobilization: A randomized, single-blind, controlled trial. Complement Ther Clin Pract. 2022 Aug;48:101580. doi: 10.1016/j.ctcp.2022.101580. Epub 2022 Apr 4. PMID 35397306